CLINICAL TRIAL: NCT02962115
Title: Development and Pilot Testing of a Clinical Informatics Lung Cancer Screening Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IRB00036974; CCCWFU 99316 (Other: Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2016-10-19; First posted 2016-11-11 (Estimated); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Decision Aid Invitation (Experimental): Electronic invitation to complete a web-based lung cancer screening decision aid
  Interventions: Behavioral: Decision Aid Invitation

INTERVENTIONS:
Behavioral: Decision Aid Invitation — electronic invitation to complete web-based decision aid

SUMMARY:
This study evaluates the feasibility of a clinical informatics system-based approach to lung cancer screening. Patients of a large academic medical center who may qualify for lung cancer screening will be sent an electronic invitation to complete an online lung cancer screening decision aid.

DETAILED DESCRIPTION:
The Center for Medicaid and Medicare Services (CMS) recently approved the use of low-dose chest CT scans for lung cancer screening in patients who meet specific criteria. However, many individuals who meet these criteria do not realize they qualify for screening. This study will determine the feasibility of using a clinical informatics approach to systematically identify potential candidates for LDCT screening, reach out to them via the patient portal, and use a web app to provide them with a personalized LDCT screening decision aid and facilitate the ordering of screening tests.

ELIGIBILITY:
Inclusion Criteria:

* Has an active patient portal account
* Scheduled to see a Wake Forest primary care provider within the next 4 weeks

Exclusion Criteria:

* Never smokers
* Current or former history of lung cancer
* Receipt of chest CT scan within last 12 months
* Need for a language interpreter
* Presence of disease predicting short life-expectancy

Ages: 55 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2016-11; Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Receipt of LDCT screening | 120 days
  Number of participants who received a low-dose chest CT

SECONDARY OUTCOMES:
Read portal invitation | 120 days
  Number of participants who read the portal invitation
Visit web decision aid | 120 days
  Number of participants who visited the study website
Complete web decision aid | 120 days
  Number of participants who complete the lung cancer screening eligibility items
Eligible for LDCT | 120 days
  Number of participants who are confirmed eligible for LDCT by the study website
Interest in LDCT screening | 120 days
  Number of participants who indicate they are interested in receiving LDCT
Appointment for LDCT visit | 120 days
  Number of participants who are scheduled for a lung cancer screening clinic visit or a LDCT exam

CONTACTS AND LOCATIONS:
Overall Officials: David P Miller, MD, MS, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dharod A, Bellinger C, Foley K, Case LD, Miller D. The Reach and Feasibility of an Interactive Lung Cancer Screening Decision Aid Delivered by Patient Portal. Appl Clin Inform. 2019 Jan;10(1):19-27. doi: 10.1055/s-0038-1676807. Epub 2019 Jan 9. PMID 30625501